CLINICAL TRIAL: NCT05035823
Title: Motor NeuroProsthesis to Restore Motor Control for the COMMAND of Digital Devices: An Early Feasibility Study (EFS) of Safety in Subjects With Severe Quadriparesis
Brief Title: COMMAND Early Feasibility Study: Implantable BCI to Control a Digital Device for People With Paralysis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Synchron Medical, Inc. (Industry)
Responsible Party: Sponsor
Organization: Synchron, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: S-02-01
Record Dates: First submitted 2021-09-01; First posted 2021-09-05 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Neurologic Disorder; Paralysis; Paralysis; Stroke; Amyotrophic Lateral Sclerosis; Muscular Dystrophies; Spinal Cord Injuries; Stroke, Lacunar; Stroke Brainstem; Cervical Spinal Cord Injury; Spinal Muscular Atrophy; Tetraplegic; Paralysis; Quadriplegia/Tetraplegia
MeSH Terms: conditions — Nervous System Diseases; Paralysis; Stroke; Amyotrophic Lateral Sclerosis; Muscular Dystrophies; Spinal Cord Injuries; Stroke, Lacunar; Brain Stem Infarctions; Muscular Atrophy, Spinal; Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single (Other): Implantation of the motor neuroprosthesis medical device.
  Interventions: Device: Motor Neuroprosthesis (MNP)

INTERVENTIONS:
Device: Motor Neuroprosthesis (MNP) — Type of implantable brain computer interface

SUMMARY:
The Synchron motor neuroprosthesis (MNP) is intended to be used in subjects with severe motor impairment, unresponsive to medical or rehabilitative therapy and a persistent functioning motor cortex. The purpose of this research is to evaluate safety and feasibility.

The MNP is a type of implantable brain computer interface which bypasses dysfunctional motor neurons. The device is designed to restore the transmission of neural signal from the cerebral cortex utilized for neuromuscular control of digital devices, resulting in a successful execution of non-mechanical digital commands.

ELIGIBILITY:
Inclusion Criteria:

1. Severe quadriparesis
2. Able to give consent
3. Appropriate candidate for neurointerventional procedure
4. Able and willing to access all clinical testing and not impeded by geographical location
5. Proficient in English
6. Have a study partner

Exclusion Criteria:

1. Active condition resulting in immunosuppression
2. Unsuitable for general anesthesia
3. Anaphylactic allergy to contrast media
4. Allergy to nickel
5. History of pulmonary embolism
6. History of recent deep vein thrombosis
7. Psychiatric or psychological disorder
8. No study partner or caregiver
9. Unable to provide evidence of COVID vaccination

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Treatment-Related Serious Adverse Events | 12 months post implant
  Number of subjects with treatment-related adverse events

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University at Buffalo Neurosurgery (UBNS), Buffalo, New York
  - Mount Sinai Health System, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Chetty N, Kacker K, Feldman AK, Yoo PE, Bennett J, Fry A, Tal I, Hardy NF, Ebrahimi S, Echavarria C, Sawyer A, Schone HR, Harel NY, Nogueira RG, Majidi S, Levy EI, Kandel A, Hill KK, Opie NL, Lacomis D, Collinger JL, Oxley TJ, Putrino DF, Weber DJ. Signal properties and stability of a chronically implanted endovascular brain computer interface. medRxiv [Preprint]. 2025 Sep 25:2025.09.19.25335897. doi: 10.1101/2025.09.19.25335897. PMID 41040697